CLINICAL TRIAL: NCT03069560
Title: Short Message System (SMS) for Caregivers of Suicidal Patients to Prevent Recidivism of Suicide Attempts
Acronym: C-SIAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C-SIAM (29.BRC.16.115)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2020-05

CONDITIONS: Prevention of the Suicide
Keywords: suicide attempt; SMS monitoring; Phone; Prevention control; tertiary healthcare
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMS (Experimental): The patients will receive from the caregiver a first SMS 48 hours after their discharge from the hospital then a total of 4 messages : 48 hours, S1, S2, and S4.
  Interventions: Device: SMS

INTERVENTIONS:
Device: SMS — SMS contact from the caregiver with patient after discharge in intervention group

SUMMARY:
Assessment of the feasibility of a monitoring device by SMS in which messages are sent by the caregiver after a suicidal act.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years of age and hospitalized;
* Survivor of a suicide attempt;
* Giving informed, dated and signed consent;
* Can be reached by mobile phone. The study is proposed to all adult suicides and to the patient's designated caregiver, meeting the inclusion criteria.

Exclusion Criteria:

* Patient whose clinical condition is incompatible with the formulation of his non-opposition.
* The patient and his / her caregiver shall not be afforded a protective justice measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the feasibility of the device by the patient according to a validated questionnaire | 6 months
  The primary endpoint is the measurement of the feasibility of the device by the patient based on a validated questionnaire. This evaluation will take place during the medical interview that will close the study participation.

SECONDARY OUTCOMES:
The questionnaire measuring the feasibility for the caregiver of such a device | 6 months
  A questionnaire will be provided to the caregiver to measure the feasibility of such a device
Questionnaires on the acceptability of patients and caregivers in relation to the use of this type of monitoring device | 6 months
  Acceptability questionnaires will be provided to patients and caregivers in relation to the use of this type of monitoring device
Qualitative analysis of messages sent to patients during the study. | 6 months
  A qualitative analysis of the messages addressed to the patients during the study will be carried out.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

REFERENCES:
- [Background] Le Moal V, Lemey C, Walter M, Berrouiguet S. Viewpoint: Toward Involvement of Caregivers in Suicide Prevention Strategies; Ethical Issues and Perspectives. Front Psychol. 2018 Dec 18;9:2457. doi: 10.3389/fpsyg.2018.02457. eCollection 2018. No abstract available. PMID 30618917